CLINICAL TRIAL: NCT01765114
Title: A Phase II Open-label, Intra-individual Controlled, Single-center Study to Investigate the Efficacy, Safety and Tolerability of a Polyethylene Glycol-formulation and the Viral Shedding in Patients Suffering From Genital Herpes
Brief Title: A Study to Investigate the Efficacy, Safety and Tolerability of PEG in Patients With Genital Herpes
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: insufficient patient recruitment
Sponsor: Devirex AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEV-PEG-02
Record Dates: First submitted 2012-12-14; First posted 2013-01-10 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Genital Herpes
MeSH Terms: conditions — Herpes Genitalis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PEG-Formulation (Experimental): PEG-Formulation, applied twice daily during the treatment period (duration: 6 months)
  Interventions: Drug: PEG-Formulation

INTERVENTIONS:
Drug: PEG-Formulation

SUMMARY:
The aim of this study is therefore to investigate the efficacy of the PEG-formulation to reduce the frequency and duration of genital herpes recurrences, to assess its safety and tolerability and to investigate its effect on shedding.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* 18 - 65 years
* Positive for HSV-1 and/or -2 (as determined by serology testing in course of study)
* Initial infection > 1 year ago
* ≥ 6 recurrences in the last year (or in the year prior to a recent prophylactic therapy)
* ≥ 2 recurrences during the six-month baseline period

Exclusion Criteria:

* Known or suspected allergy or intolerability to PEG
* Prophylactic antiviral drugs, virostatic agents, cytostatics, immunomodulatory drugs and steroids within less than 14 days prior to baseline period, or plan to take such drugs during the trial
* Pregnancy and/or breast-feeding
* History of malignant diseases (described in chapter 7.2)
* Known or suspected non-compliance to study protocol
* Participation in another investigational drug study in the last 30 days prior to baseline period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change of number of genital herpes recurrences during the treatment period as compared to the baseline period. | Baseline and Treatment period (6 months each).
  The number of genital herpes recurrences will be counted during the baseline period (6 months) and during the treatment period (6 months) and then be compared.

SECONDARY OUTCOMES:
The safety of the PEG-formulation via reporting of AEs. | Baseline and Treatment period (6 months each).

OTHER OUTCOMES:
The frequency of days with viral shedding which will be analysed by quantitative PCR. | Baseline and Treatment period (6 months each).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kuendig, MD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland